CLINICAL TRIAL: NCT00020748
Title: A Phase I Study of Epirubicin in Combination With Irinotecan in Patients With Advanced Cancer
Brief Title: Epirubicin Plus Irinotecan in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John Marshall, MD, Georgetown University
Purpose: Treatment
Other Study IDs: CDR0000068710; P30CA051008 (NIH); GUMC-00191; GUMC-072000-001; NCI-G01-1956
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2005-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Epirubicin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epirubicin hydrochloride
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of epirubicin plus irinotecan in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxicity and maximum tolerated dose of epirubicin and irinotecan in patients with advanced cancer.
* Determine the objective antitumor responses in patients treated with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive irinotecan IV over 1 hour followed by epirubicin IV over 5 minutes on days 1 and 8. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Sequential dose escalation of epirubicin is followed by sequential dose escalation of irinotecan. Cohorts of 3-6 patients receive escalating doses of epirubicin and irinotecan until the maximum tolerated dose (MTD) of each is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically documented incurable malignancy for which there is no beneficial standard therapy

  * Locally unresectable or metastatic disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 8 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.2 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 2 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* Ejection fraction at least 50% by MUGA scan
* No congestive heart failure

Other:

* Maintaining a reasonable state of nutrition
* No frequent vomiting or severe anorexia
* No weight loss greater than 10% of current body weight within the past 4 weeks
* No other concurrent medical illness that would preclude study
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* Prior doxorubicin allowed if cumulative dose no greater than 240 mg/m2

Endocrine therapy:

* Not specified

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* Recovered from prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L. Marshall, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (1):
- Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia, United States